CLINICAL TRIAL: NCT04244825
Title: A Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate Pharmacodynamics, Pharmacokinetics, and Safety of BLD-2660 Administered Orally in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Safety, Pharmacodynamics, and Pharmacokinetics of Orally Administered BLD-2660 in Subjects With IPF
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to concerns for patient safety during COVID-19 crisis
Sponsor: Blade Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-2660-203
Record Dates: First submitted 2020-01-03; First posted 2020-01-28 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1a BLD-2660 (Experimental): 900 mg (6 x 150 mg capsules) BID
  Interventions: Drug: BLD-2660
- Cohort 1b BLD-2660 (Experimental): 900 mg (6 x 150 mg capsules) BID (Optional)
  Interventions: Drug: BLD-2660
- Cohort 2 BLD-2660 (Experimental): 600 mg (4 x 150 mg capsules) BID
  Interventions: Drug: BLD-2660
- Cohort 3 BLD-2660 (Experimental): 300 mg (2 x 150 mg capsules) BID
  Interventions: Drug: BLD-2660
- Cohort 1a Placebo (Placebo Comparator): 900 mg (6 x 150 mg capsules) BID
  Interventions: Drug: Control: Placebo
- Cohort 1b Placebo (Placebo Comparator): 900 mg (6 x 150 mg capsules) BID (Optional)
  Interventions: Drug: Control: Placebo
- Cohort 2 Placebo (Placebo Comparator): 600 mg (4 x 150 mg capsules) BID
  Interventions: Drug: Control: Placebo
- Cohort 3 Placebo (Placebo Comparator): 300 mg (2 x 150 mg capsules) BID
  Interventions: Drug: Control: Placebo

INTERVENTIONS:
Drug: BLD-2660 — BLD-2660 - 150 mg capsules '00' size (PO) BID
  Arms: Cohort 1a BLD-2660; Cohort 1b BLD-2660; Cohort 2 BLD-2660; Cohort 3 BLD-2660
Drug: Control: Placebo — Placebo - 150 mg capsules '00' size (PO) BID
  Arms: Cohort 1a Placebo; Cohort 1b Placebo; Cohort 2 Placebo; Cohort 3 Placebo

SUMMARY:
A Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate Pharmacodynamics, Pharmacokinetics, and Safety of BLD-2660 Administered Orally in Subjects with Idiopathic Pulmonary Fibrosis

DETAILED DESCRIPTION:
This is a Phase 2a, double-blind, placebo-controlled, multicentre, adaptive design study of BLD-2660 in subjects with IPF. The study will include a Screening period, a Treatment period, and a Follow-up period. Data on PK, PD, and biomarker activity will be observed.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this study, each subject must fulfill the following inclusion criteria within 20 days prior to Randomization on Day 1:

Age and Gender

1. Male subjects 45 years of age and over, or female subjects 50 years of age and over, at the time of signing the informed consent.

   Diagnosis and disease characteristics
2. Subjects with diagnosis of IPF as defined by the American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of Idiopathic Interstitial Pneumonia.
3. Forced vital capacity (FVC) >45% predicted and diffusing capacity of the lung for carbon monoxide (DLCO) >30% predicted.
4. Alanine aminotransferase (ALT) within normal limit (WNL).
5. Aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤1.2× upper limit of normal (ULN).
6. Total bilirubin ≤ULN (isolated bilirubinemia ≤2× ULN is acceptable if direct bilirubin to total bilirubin ratio <0.35).
7. Body mass index (BMI) up to 35 kg/m2 inclusive. Reproductive Considerations Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
8. All subjects (male or female) who are of childbearing potential must agree to use highly effective contraception during the study.
9. Male subjects and female partners of male subjects must continue to use highly effective contraception for 90 days after the last dose of study drug (see Medicines and Healthcare products Regulatory Agency, 2019 for further guidance regarding highly effective contraception). Male subjects must agree not to donate sperm for 90 days after last dose of study drug.
10. Female subjects and male partners of female subjects must continue to use highly effective contraception for 60 days after the last dose of study drug. Female subjects should not donate oocytes during this time.
11. Female subjects of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day (-1). Women of childbearing potential (WOCBP) must agree to undergo pregnancy testing at regular intervals throughout the study.
12. Female subjects not of childbearing potential as defined by being postmenopausal (with cessation of regular menstrual periods for at least 1 year), confirmed by follicle stimulating hormone (FSH) level, or be surgically sterile.

    Informed Consent
13. Subjects must provide signed informed consent prior to study entry and have the ability and willingness to attend and comply with the necessary visits at the study site.

Exclusion Criteria:

To be eligible for inclusion into this study, each subject must violate none of the following exclusion criteria within 20 days prior to Randomisation on Day 1.

Medical Conditions

1. Recent (less than 6 weeks) significant wound (in the opinion of the Investigator), or presence of an ongoing non-healing skin wound or ulcer.
2. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the subject will complete the study per protocol.
3. Active infection (diagnosed or suspected) or history of recurrent infections, including but is not limited to, bronchitis, pneumonia, sinusitis, urinary tract infection, cellulitis or chronic ongoing infectious disease within 4 weeks prior to first dose of study drug. Note: Rescreening will be permitted after 28 days if an infection leads to screening failure.
4. Active malignancy and/or history of malignancy in the past 5 years, except for non-melanoma skin cancer, carcinoma in situ of the breast that has been successfully treated, carcinoma in situ of the cervix that has been successfully treated, early stage, untreated prostate cancer, or prostate cancer with completion of treatment >2 years prior to Screening.
5. Extensive chronic obstructive pulmonary disease (where extent of emphysema >extent of fibrosis on computerised tomography (CT) scan or FEV1: FVC ratio <0.65).
6. Other explanation for lung fibrosis, including but not limited to radiation, sarcoidosis, bronchiolitis obliterans organizing pneumonia, collagen vascular disease, hypersensitivity pneumonitis, etc.
7. IPF exacerbation within last 60 days.
8. A history or current evidence of any medical condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subjects' participation for the full duration of the study, or is not in the best interest of the subjects to participate, in the opinion of the Investigator.

   Diagnostic Assessments
9. Positivity for Human Immunodeficiency Virus (HIV) antibody (HIV-1 and/or HIV-2) and/or HIV-1 p24 antigen.
10. Positivity for Hepatitis C virus antibody (HCV Ab or anti-HCV) and/or Hepatitis B surface antigen (HBsAg).
11. Absolute neutrophil count <1700/µL.
12. Significant hypoxia, requiring >2 L/min oxygen to maintain a resting oxygen saturation >89%.
13. Poor exercise tolerance.
14. Serum troponin I level >ULN.

    Prior/Concomitant Therapy
15. Use of anticoagulants that prolong Prothrombin time (PT)/International normalised ratio (INR).
16. Use of anticoagulants within 2 days of Day (-1) (bronchoscopy). Note: The subjects who cannot discontinue the anticoagulants within 2 days of Day (-1) bronchoscopy will be excluded.
17. Treatment with any anti-fibrotic therapy (pirfenidone or nintedanib) within 30 days of Screening.
18. Immunosuppressive therapy within 3 months prior to first dose of study drug (unless for non-IPF indication).
19. Use of oral steroids >10 mg/day (or prednisolone equivalent). Note: If the subject is on steroid dose equivalent to 10 mg/day prednisone or more, the Investigator may decide if the tapering down to the dose of 10 mg/day prednisone is possible and safe.
20. Start of new biologic or change in biologic dose within 24 weeks prior to Day 1.
21. Cyclophosphamide within 6 months prior to the first dose of study drug (unless for other indication).

    Prior/Concurrent Clinical Study Experience
22. Administration of another investigational product, investigational device, or approved therapy for investigational use within 30 days prior to the first study drug administration, or five half-lives, whichever is longer.

    Other Exclusions
23. Blood donation or significant blood loss within 60 days prior to the first study drug administration.
24. Plasma donation within 7 days prior to the first study drug administration.
25. Female subjects who are pregnant or breastfeeding.
26. History or presence of alcohol or drug abuse (including recreational marijuana use) within the 2 year prior to the first study drug administration, and unwillingness to be totally abstinent during the dosing period.
27. Active smoker, smoking history or vaping within 4 weeks prior to the first dose of study drug. Subjects only using Nicotine replacement therapy (NRT) may be allowed per discretion of the Investigator.
28. Subjects with an allergy to BLD-2660 or inactive components of BLD-2660.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Observed changes in ILK from baseline | 58 days
  Change in RLU of BAL fluid analyzed by ILK-targeting ELISA assay. Analysis of difference in RLU correlates to change in cellular ILK from baseline.
Observed changes in spectrin from baseline | 58 days
  Change in RLU of BAL fluid analyzed by spectrin-targeting ELISA assay. Analysis of difference in RLU correlates to change in cellular spectrin from baseline.
Observed changes in ezrin from baseline | 58 days
  Change in RLU of BAL fluid analyzed by ezrin-targeting ELISA assay. Analysis of difference in RLU correlates to change in cellular ezrin from baseline.
Observed changes in S100A9 from baseline | 58 days
  Change in RLU of BAL fluid analyzed by S100A9-targeting ELISA assay. Analysis of difference in RLU correlates to change in cellular S100A9 from baseline.

SECONDARY OUTCOMES:
Area under the drug concentration-time curve from time zero to the last measurable concentration (AUC0-last) | 58 days
  Measured by plasma concentration
AUC from time 0 to infinity (AUC0-inf) | 58 days
  Measured by plasma concentration
Maximum observed drug concentration (Cmax) | 58 days
  Measured by plasma concentration
Time of the maximum drug concentration (Tmax) | 58 days
  Measured by plasma concentration
Incidence of Treatment-Emergent Adverse Events as assessed by PI and SMC | 58 days
  AEs will be assessed by determining the incidence, severity, and dose relationship of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Blade Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No